CLINICAL TRIAL: NCT03547102
Title: Effect of Cherry Concentrate on Brain Activation and Perfusion in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 115229/02
Record Dates: First submitted 2016-12-02; First posted 2018-06-06 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cherry concentrate (Active Comparator): 8 weeks supplementation with montmorency cherry concentrate
  Interventions: Dietary Supplement: Cherry concentrate
- Placebo concentrate (Placebo Comparator): 8 weeks supplementation with placebo isoenergetic cherry concentrate
  Interventions: Dietary Supplement: Placebo concentrate

INTERVENTIONS:
Dietary Supplement: Cherry concentrate
  Arms: Cherry concentrate
Dietary Supplement: Placebo concentrate
  Arms: Placebo concentrate

SUMMARY:
Effect of 8 weeks of cherry concentrate supplementation on cognitive function and brain perfusion in healthy older adults

DETAILED DESCRIPTION:
The investigators will perform a double blind, randomised controlled study to determine whether cherry polyphenols improve peripheral vascular function and cerebral perfusion resulting in improved task related brain activation and cognitive function. 30 healthy elderly men and women 60-85y years will be recruited to complete 8-week supplementation with MC concentrate or an isoenergetic cherry placebo concentrate. Participants will be pair matched for age, sex, and cognitive function (Adenbrooke's Cognitive Examination III, ACE-III) and then randomised using a sealed envelope system to receive either placebo or cherry.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive consuming 5 or less portions of fruit per day Addenbrookes cognitive examination III score >88

Exclusion Criteria:

* physically active consuming more than 5 portions of fruit per day Addenbrookes cognitive examination III score <88 Contraindications for MRI

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Brain perfusion | Change from baseline to 8 weeks supplementation
  Arterial spin labelling using MRI, measure will be reported as ml/min

SECONDARY OUTCOMES:
Cognitive function | Change from baseline to 8 weeks supplementation
  Battery of cognitive function tasks assessing executive function, global cognitive function score will be reported
Brain activation (fMRI) | Change from baseline to 8 weeks supplementation
  fMRI using a hippocampal biased task
Plasma nitrite concentration | Change from baseline to 8 weeks supplementation
  Plasma sample analysed via chemiluminescence technique

CONTACTS AND LOCATIONS:
Overall Officials: Joanna L Bowtell, PhD, Principal Investigator — University of Exeter

IPD SHARING:
Plan to Share IPD: No